CLINICAL TRIAL: NCT03811639
Title: ABLation-induced Changes in Cardiac Autonomic Nervous System in Patients With Atrial Fibrillation: Radiofrequency Versus Cryoballoon Techniques. The ABLANSAF Study.
Brief Title: Changes in Cardiac Autonomic Nervous System Following Atrial Fibrillation Ablation.
Acronym: ABLANSAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, head of Electrophysiology Department, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65/PB/2015
Record Dates: First submitted 2018-12-29; First posted 2019-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: ablation, atrial fibrillation, autonomic nervous system
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Comparison of changes in autonomic heart regulation caused by radio-frequency ablation and cryoballoon ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF ablation (Active Comparator): Patients treated with point-by-point radio-frequency ablation
  Interventions: Procedure: Radio-frequency ablation
- Cryoballoon ablation (Experimental): Patients treated with cryoballoon ablation
  Interventions: Procedure: Cryoballoon ablation

INTERVENTIONS:
Procedure: Radio-frequency ablation — Ablation for atrial fibrillation
  Arms: RF ablation
Procedure: Cryoballoon ablation — Ablation for atrial fibrillation
  Arms: Cryoballoon ablation

SUMMARY:
Aim. To compare changes in cardiac autonomic tone caused by radio-frequency versus cryoballoon ablation and to assess their value in predicting the outcome.

Study group. In this prospective randomized study 126 consecutive patients with paroxysmal AF undergoing first ablation of AF using radio-frequency (RF) or cryoballoon (CB) technique will be recruited. Patients will undergo several ECG and autonomic tests before and after the procedure. The follow-up will last one year.

Measurements:

1. Standard 12-lead ECG a day before and 1-2 days after the procedure will be performed. The SR and P wave duration as well as the difference (∆) in SR and P wave duration before and after ablation will be analyzed.
2. A 24-hour Holter ECG will be performed at baseline (1-2 days before ablation) and 7-day Holter ECG will be performed 3, 6 and 12 months after the procedure. Minimal, maximal and mean heart rate (HR) as well as HRV parameters will be analyzed. The differences (∆) in these variables between baseline and post-ablation Holter ECG recordings will be analyzed.
3. Autonomic parameters (HR, HRV parameters and baroreceptor reflex sensitivity as well as hemodynamic parameters (stroke volume (SV), cardiac output (CO), total peripheral resistance (TPR)) will be also examined before and after orthostatic stress. This will be performed using tilt table test and non-invasive measurement of autonomic and hemodynamic parameters before and shortly after (1-3 days) the procedure.
4. Quality of life will be assessed using the AFSS scale and EHRA scale at baseline and 3, 6 and 12 months after ablation.
5. Follow-up will last 12 months. Efficacy of ablation will be assessed during outpatients visits and using 7-day Holter ECG recordings 3, 6 and 12 months after the procedure. The analyzed outcomes will include symptomatic recurrences of AF, hospitalizations due to AF, redo procedures i occurrence of asymptomatic AF on Holter ECG monitoring.
6. All the above listed parameters and ablation efficacy will be compared between the RF and CB groups.

Anticipated results.

1. Ablation significantly effects the parameters of cardiac autonomic control
2. These effects are more pronounced in the CB group compared with the RF group
3. Changes in autonomic indices have value in predicting ablation efficacy in both analyzed groups.

DETAILED DESCRIPTION:
ABLation-induced changes in cardiac Autonomic Nervous System in patients with Atrial Fibrillation: radiofrequency versus cryoballoon techniques (the ABLANSAF study).

Introduction. The primary goal of ablation for atrial fibrillation (AF) is pulmonary vein isolation (PVI). The second mechanism of action of ablation is modification of cardiac autonomic tone by ablation of atrial ganglionated plexi, mainly of their parasympathetic component. Data in literature concerning this topic is scares. A few studies showed that ablation-induced changes in heart rate variability (HRV) or sinus rate (SR) predict the outcome. However, these data are preliminary and have not yet been included into clinical practice. Moreover, whether these effects depend on the technique used - radio-frequency (RF) ablation or cryoballoon (CB) ablation, has not yet been examined.

Aim. To compare the changes in cardiac autonomic tone caused by RF versus CB ablation and to assess their value in predicting the outcome after the procedure.

Hypothesis. We hypothesised that both techniques cause significant changes in cardiac autonomic innervation, however, these changes are significantly more pronounced following CB rather than RF ablation.

Methods. Study group. In this prospective randomised study 126 consecutive patients with paroxysmal AF undergoing first ablation of AF using RF or CB technique will be recruited. Patients will undergo several ECG and autonomic tests before and after the procedure. The follow-up will last one year.

Ablation The RF and CB ablation will be performed using standard approach. A patient will be randomly selected to RF or CB ablation. The only parameter influencing randomisation will be the presence of the common trunk of the left PV (visualised by computed tomography or rotational angiography) which is regarded as relative contraindication to CB because of anatomical difficulties in the positioning of balloon. In such cases the decision as to the type of procedure will be left to the discretion of the operator.

The CB PVI will be conducted in standard manner. Briefly, after injection of local anesthetic, both femoral veins is punctured. One long sheath (8.5 F Swartz, St. Jude, Saint Paul, USA) to cross interatrial septum is inserted in the right femoral vein. Another two short sheaths were inserted in the left femoral vein for the intracardiac echocardiographic probe (8 or 10 Fr Acunav, Acuson, Siemens, Berlin) and diagnostic catheter introduced into the coronary sinus. After crossing the septum and introducing guidewire into the left superior pulmonary vein (LSPV), long sheath is replaced with steerable sheath (14 F., Flexcath, Medtronic, Minneapolis, USA) and CB (28 mm, second generation) is introduced into the left atrium. Next, the Achieve (20 mm diameter) mapping catheter, (Medtronic, Milwaukee, USA) is placed in the LSPV ostium, CB inflated and contrast injected to confirm proper occlusion of LSPV. When PVI is achieved during first freezing lasting 180 - 240 sec and confirmed by PV potentials (PVP) disappearance within 60 seconds by recordings from the Achieve catheter, no second cryoapplication is performed. In case of incomplete occlusion, persistence or very late disappearance of PVP, suboptimal temperatures achieved (less than -36C) or very short thawing time, CB is repositioned and another cryo-application is delivered. Next, CB-PVI of the left inferior pulmonary vein (LIPV), right superior pulmonary vein (RSPV) and right inferior pulmonary vein (RIPV) is performed. Pacing of the right phrenic nerve is performed during CB of the right veins to avoid phrenic nerve palsy.

The RF ablation is performed in a standard manner using 3-D electro-anatomical system CARTO-3 (Biosense Webster, USA) and Smarttouch ablation catheter. Two separate transseptal punctures are performed under intracardiac echocardiography guidance. After reconstruction of the left atrial geometry using merging of the computed tomography or rotational angiography image with the CARTO map, the point-by-point PVI of each vein is performed. The ablation index is used to ensure the quality of RF applications. The Lasso circular catheter (Biosense Webster, USA) is used to assess PVI and diagnostic catheter placed in the coronary sinus is used for pacing manoeuvres.

Measurements:

1. Standard 12-lead ECG a day before and 1-2 days after the procedure will be performed. The SR and P wave duration as well as the difference (∆) in SR and P wave duration before and after ablation will be analysed.
2. A 24-hour Holter ECG will be performed at baseline (1-2 days before ablation) and 7-day Holter ECG will be performed 3, 6 and 12 months after the procedure. Minimal, maximal and mean heart rate (HR) as well as time-domain HRV parameters (SDNN, SDANN, pNN50, rMSSD) and frequency-domain HRV indices (LF, HF, LF/HF) will be analysed. The differences (∆) in these variables between baseline and post-ablation Holter ECG recordings will be analysed.
3. Autonomic parameters (HR, frequency-domain HRV parameters and baro-reflex sensitivity (BRS) using sequential method) as well as hemodynamic parameters (stroke volume (SV), cardiac output (CO), total peripheral resistance (TPR)) will be also examined before and after orthostatic stress. This will be performed using tilt table test (70 degrees) and non-invasive measurement of autonomic and hemodynamic parameters (cardiac impedance method) using the Task Force system, before (1-2 days) and shortly after (1-3 days) the procedure. The 5-min ECG recordings will be used to calculate the values of autonomic and haemodynamic parameters. Also ∆ of these parameters will be computed. The values measured before and after ablation, before and after tilt testing as well ∆ will be compared.
4. Quality of life will be assessed using the AFSS scale and EHRA scale at baseline and 3, 6 and 12 months after ablation.
5. Follow-up will last 12 months. Efficacy of ablation will be assessed during outpatients visits and using 7-day Holter ECG recordings 3, 6 and 12 months after the procedure. The analysed outcomes will include symptomatic recurrences of AF, hospitalisations due to AF, redo procedures i occurrence of asymptomatic AF on Holter ECG monitoring. Efficacy of the procedure will be assessed and defined as (1) complete efficacy - no symptoms attributed to AF and no AF on Holter ECG monitoring; (2) symptomatic efficacy - no symptoms attributed to AF but AF episodes > 30 sec recorded on Holter ECG monitoring; (3) partial efficacy - recurrences of symptomatic AF, however, of lower intensity, defined as improvement of at least 1 degree in the EHRA scale and improvement in the AFSS scale; and (4) no effects - no change in symptoms compared with the pre-ablation periods.
6. All the above listed parameters and ablation efficacy will be compared between the RF and CB groups.

Statistical analysis. The results will be presented as mean±SD (normally distributed variables) or median values (not normally distributed variables). The changes between baseline and parameters obtained after ablation as well as before and after tilt testing will be performed using paired two-tailed Student t-test, Mann-Whitney or ANOVA tests where appropriate. The results obtained in the RF versus CB groups will be compared using unpaired Student t-test. The predictive value of examined parameters in identifying responders to ablation will be assessed using the ROC curves and by computing sensitivity, specificity, positive and negative predictive value. Multivariate analysis will be performed to identify parameters independently associated with ablation efficacy. A p value < 0.05 will be considered significant.

The estimated number of patients sufficient to detect significant difference between the RF and CB groups is 126 based on the assumption that ablation-induced changes in cardiac autonomic parameters will differ between the RF and CB groups by 20% (alfa error = 0.05 and beta error = 0.2) Anticipated results.

1. Ablation significantly effects the parameters of cardiac autonomic control
2. These effects are more pronounced in the CB group compared with the RF group
3. Changes in autonomic indices have value in predicting ablation efficacy in both analysed groups.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal AF
* First AF ablation
* Sinus rhythm before and after the procedure at the time of ECG and tilt table testing.
* No change in medication affecting cardiac autonomic nervous system before and after ablation.
* Obtained written informed consent to participate in the study.

Exclusion Criteria:

* Any of inclusion criterion not met
* Pacing system implanted
* Additional ablation to PVI like cavo-tricuspid isthmus ablation or linear lesions in the left atrium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate-induced changes in the RF and CB groups. | 1-2 days before and 2-3 days after ablation heart rate will be recorded
  The baseline and tilt-induced heart rate (beats/min) measured before and after ablation will be compared between the RF and CB groups
Heart rate variability (SDNN)-induced changes in the RF and CB groups. | 1-2 days before and 2-3 days after ablation SDNN parameter will be recorded
  The baseline and tilt-induced heart rate variability (SDNN) (msec) measured before and after ablation will be compared between the RF and CB groups
Baroreflex sensitivity-induced changes in the RF and CB groups. | 1-2 days before and 2-3 days after ablation baroreflex sensitivity will be recorded
  The baseline and tilt-induced baroreflex sensitivity (msec/mmHg) measured before and after ablation will be compared between the RF and CB groups

SECONDARY OUTCOMES:
Efficacy of RF versus CB ablation (ECG symptomatic AF recurrences) | One year
  Efficacy of RF versus CB ablation will be compared using repetitive Holter ECG monitoring and documented on ECG symptomatic AF recurrences during one year follow-up
Ablation-induced changes in heart rate predicting ablation efficacy | One year
  Ablation-induced change in heart rate (beats/min) will be analyzed as a predictor of ablation efficacy during one-year follow-up
Ablation-induced changes in heart rate variability predicting ablation efficacy | One year
  Ablation-induced change in heart rate variability (SDNN) (msec) will be analyzed as a predictor of ablation efficacy during one-year follow-up
Ablation-induced changes in baroreflex sensitivity predicting ablation efficacy | One year
  Ablation-induced change in baroreflex sensitivity (msec/mmHg) will be analyzed as a predictor of ablation efficacy during one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulakowski, MD, Study Chair — Postgraduate Medical School, Grochowski Hospital
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
All study data will be available to other researchers or reviewers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During the study and up to 5 years after study termination
Access Criteria: Data will be available for researchers who are interested in this field and to reviewers if they ask for data during reviewing process

REFERENCES:
- [Background] Hsieh MH, Chiou CW, Wen ZC, Wu CH, Tai CT, Tsai CF, Ding YA, Chang MS, Chen SA. Alterations of heart rate variability after radiofrequency catheter ablation of focal atrial fibrillation originating from pulmonary veins. Circulation. 1999 Nov 30;100(22):2237-43. doi: 10.1161/01.cir.100.22.2237. PMID 10577997
- [Result] Pappone C, Santinelli V, Manguso F, Vicedomini G, Gugliotta F, Augello G, Mazzone P, Tortoriello V, Landoni G, Zangrillo A, Lang C, Tomita T, Mesas C, Mastella E, Alfieri O. Pulmonary vein denervation enhances long-term benefit after circumferential ablation for paroxysmal atrial fibrillation. Circulation. 2004 Jan 27;109(3):327-34. doi: 10.1161/01.CIR.0000112641.16340.C7. Epub 2004 Jan 5. PMID 14707026
- [Result] Yamada T, Yoshida N, Murakami Y, Okada T, Yoshida Y, Muto M, Inden Y, Murohara T. Vagal modification can be a valid predictor of late recurrence of paroxysmal atrial fibrillation independent of the pulmonary vein isolation technique. Circ J. 2009 Sep;73(9):1606-11. doi: 10.1253/circj.cj-09-0158. Epub 2009 Jul 17. PMID 19609042
- [Result] Yamada T, Yoshida N, Murakami Y, Okada T, Yoshida Y, Muto M, Inden Y, Murohara T. The difference in autonomic denervation and its effect on atrial fibrillation recurrence between the standard segmental and circumferential pulmonary vein isolation techniques. Europace. 2009 Dec;11(12):1612-9. doi: 10.1093/europace/eup330. Epub 2009 Oct 29. PMID 19875397
- [Result] Yamaguchi Y, Kumagai K, Nakashima H, Saku K. Long-term effects of box isolation on sympathovagal balance in atrial fibrillation. Circ J. 2010 Jun;74(6):1096-103. doi: 10.1253/circj.cj-09-0899. Epub 2010 May 8. PMID 20467150
- [Result] Oswald H, Klein G, Koenig T, Luesebrink U, Duncker D, Gardiwal A. Cryoballoon pulmonary vein isolation temporarily modulates the intrinsic cardiac autonomic nervous system. J Interv Card Electrophysiol. 2010 Oct;29(1):57-62. doi: 10.1007/s10840-010-9491-7. Epub 2010 Jun 16. PMID 20556498
- [Result] Lim PB, Malcolme-Lawes LC, Stuber T, Koa-Wing M, Wright IJ, Tillin T, Sutton R, Davies DW, Peters NS, Francis DP, Kanagaratnam P. Feasibility of multiple short, 40-s, intra-procedural ECG recordings to detect immediate changes in heart rate variability during catheter ablation for arrhythmias. J Interv Card Electrophysiol. 2011 Nov;32(2):163-71. doi: 10.1007/s10840-011-9580-2. Epub 2011 Jun 7. PMID 21647641
- [Result] Wang K, Chang D, Chu Z, Yang Y, Gao L, Zhang S, Xia Y, Dong Y, Yin X, Cong P, Jia J. Denervation as a common mechanism underlying different pulmonary vein isolation strategies for paroxysmal atrial fibrillation: evidenced by heart rate variability after ablation. ScientificWorldJournal. 2013 Aug 24;2013:569564. doi: 10.1155/2013/569564. eCollection 2013. PMID 24058286
- [Result] Seaborn GE, Todd K, Michael KA, Baranchuk A, Abdollah H, Simpson CS, Akl SG, Redfearn DP. Heart rate variability and procedural outcome in catheter ablation for atrial fibrillation. Ann Noninvasive Electrocardiol. 2014 Jan;19(1):23-33. doi: 10.1111/anec.12098. Epub 2013 Sep 24. PMID 24112475
- [Result] Kang KW, Kim TH, Park J, Uhm JS, Joung B, Hwang C, Lee MH, Pak HN. Long-term changes in heart rate variability after radiofrequency catheter ablation for atrial fibrillation: 1-year follow-up study with irrigation tip catheter. J Cardiovasc Electrophysiol. 2014 Jul;25(7):693-700. doi: 10.1111/jce.12398. Epub 2014 Mar 28. PMID 24575794
- [Result] Mori H, Kato R, Ikeda Y, Goto K, Tanaka S, Asano S, Shiki Y, Nagase T, Iwanaga S, Nishimura S, Muramatsu T, Matsumoto K. Analysis of the heart rate variability during cryoballoon ablation of atrial fibrillation. Europace. 2018 Aug 1;20(8):1259-1267. doi: 10.1093/europace/eux225. PMID 29016780
- [Result] Yu HT, Kim TH, Uhm JS, Kim JY, Joung B, Lee MH, Pak HN. Prognosis of high sinus heart rate after catheter ablation for atrial fibrillation. Europace. 2017 Jul 1;19(7):1132-1139. doi: 10.1093/europace/euw142. PMID 27256421